CLINICAL TRIAL: NCT06989229
Title: Prospective Study on the Impact of Perioperative Nutritional Care in Patients Undergoing Total Knee and Hip Arthroplasty on Postoperative Outcomes
Brief Title: The Effect of Perioperative Nutritional Care on Recovery After Knee and Hip Replacement Surgery
Status: Recruiting | Type: Observational
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Principal Investigator, Vasileios Apostolopoulos, Orthopedic Surgeon, St. Anne's University Hospital Brno, Czech Republic
Other Study IDs: 7V/2025
Record Dates: First submitted 2025-05-13; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Outcomes; Postoperative Complications; Length of Hospital Stay
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study will assess the impact of standardized perioperative nutritional care on postoperative outcomes in patients undergoing elective total hip (THA) or knee arthroplasty (TKA) at the First Department of Orthopaedic Surgery, St. Anne's University Hospital in Brno. The protocol includes preoperative patient education, nutritional risk screening, and carbohydrate loading up to two hours before anesthesia, followed by early postoperative refeeding.

Data collection will include demographic and surgical variables, nutritional status, carbohydrate intake, and the occurrence of intra- and postoperative complications, including infection and delayed wound healing.

As perioperative nutritional care is part of routine clinical practice, the study requires no additional interventions or resources. Results will provide evidence on the effectiveness of structured nutritional support in enhancing recovery and reducing complications after joint replacement surgery.

DETAILED DESCRIPTION:
At the First Department of Orthopaedics of St. Anne's University Hospital in Brno, nutritional intervention is an established and integral part of care for patients undergoing total knee and hip arthroplasty. As part of long-term preoperative preparation, emphasis is placed on patient education and the optimization of their nutritional status even before hospital admission. Education on the importance of proper nutrition is provided through the Patient Academy, where preoperative nutritional risk is also assessed. In patients identified as being at nutritional risk, targeted efforts are made to improve their nutritional status.

Preoperative fasting is an outdated method of preparing for surgical stress and can negatively affect the overall recovery process. Therefore, our clinic focuses on eliminating fasting by using carbohydrate loading, allowing patients to consume a carbohydrate drink up to two hours before the induction of anesthesia. After surgery, early refeeding is consistently applied, which supports faster recovery and reduces the risk of complications.

The aim of this study is to investigate the impact of specialized perioperative nutritional care on postoperative outcomes, with the primary objective being to assess the occurrence of postoperative complications and the length of hospital stay. For this purpose, a wide range of clinical data will be collected and analyzed, including patient age, type of surgery, BMI (body mass index), preoperative nutritional risk, amount of carbohydrate drink consumed (including taste rating), occurrence of intraoperative complications-especially aspiration-and postoperative complications such as infections and wound healing issues, as well as length of hospitalization. Data will be securely stored in the REDCap (Research Electronic Data Capture) system.

The research project will be conducted at the 1st Department of Orthopaedics of St. Anne's University Hospital in Brno (sponsor), and will include all patients undergoing elective total hip (THA) or knee (TKA) arthroplasty for whom carbohydrate loading is indicated. The implementation of the study will not incur any additional costs, as preoperative nutritional care is already a standard and established part of routine care for patients undergoing elective joint replacements. The study will provide important insights into the effectiveness of specialized nutritional care in the perioperative period and its impact on overall postoperative outcomes.

Preoperative Fasting and Nutritional Preparation Preoperative fasting is considered an unsuitable approach to preparing for surgical stress. Therefore, international societies such as ESA - European Society of Anaesthesiology and Intensive Care, ERAS - Enhanced Recovery After Surgery and ESPEN - European Society for Clinical Nutrition and Metabolism recommend minimizing fasting periods to support improved postoperative recovery.

Oral Intake Before Surgery The final meal before surgery is dinner, including a late-night snack, which is part of the low-residue diet provided by the dietary system at St. Anne's University Hospital in Brno. On the day before surgery, patients are routinely prescribed a low-residue diet (Diet No. 5) with possible modifications (5MM, 5ML, 5BML, 0/5). Patients with diabetes mellitus or impaired glucose tolerance are prescribed a diabetic low-residue diet (Diet No. 9/5), with appropriate modifications (9/5MM, 9/5ML, 90/5). Diet orders are entered into the hospital information system (NIS-SP) no later than 14:00 on the day prior to surgery.

Carbohydrate Loading

Carbohydrate loading is prescribed by the admitting physician in the orthopedic outpatient clinic based on the following criteria:

Indications:

Elective surgical procedure

Total knee or hip arthroplasty (TKA, THA)

Age ≥ 18 years

Contraindications:

Diabetes mellitus requiring insulin therapy

Carbohydrate drink schedule:

Preoperative day: PreOp 200 ml at 18:00

Day of surgery: PreOp 200 ml no later than 2 hours before anesthesia

In cases of gastrointestinal motility disorders or significant hiatal hernia, the preoperative fasting window is extended up to 4 hours. If the patient is scheduled first on the operating list, the morning dose is administered postoperatively in the ICU - Intensive Care Unit. The PreOp drink is stored refrigerated on the ward for improved taste.

Carbohydrate loading is monitored using a dedicated form ("Preoperative Preparation - Carbohydrate Loading"), given to the patient during education. The form includes patient identification, instructions, a checklist calendar, and a taste rating section. Patients record the volume consumed, which is verified by nursing staff. The completed form is placed in the patient's medical record and, after ICU discharge, stored in the departmental file accessible to the clinical dietitian.

Mechanical Bowel Preparation

Patients do not undergo mechanical bowel preparation if:

They had a bowel movement on the day before surgery

They have regular bowel habits and no chronic constipation

If necessary, a glycerin suppository is the first-line method. If ineffective, more invasive methods such as a rectal enema may be considered.

Oral Intake After Surgery Oral intake is resumed immediately postoperatively once the patient regains consciousness. The first postoperative meal is dinner, including a late-night snack, which follows the hospital's low-residue diet protocol.

On the day of surgery, patients are prescribed a low-residue diet (Diet No. 5) with applicable modifications (5MM, 5ML, 5BML, 0/5). Diabetic patients or those with impaired glucose tolerance receive a diabetic low-residue diet (Diet No. 9/5) with appropriate modifications (9/5MM, 9/5ML, 90/5).

ELIGIBILITY:
Inclusion Criteria:

Elective total hip replacement Elective total knee replacement

Exclusion Criteria:

Hip fracture Diabetes mellitus 1 Insulinotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients to undergo elective total hip and knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Complications | 2 weeks postoperatively
  Measurement: Number and type of complications documented in the patient's medical records during hospitalization and up to discharge, including infections, aspiration, and other clinical events.

SECONDARY OUTCOMES:
Length of Hospital Stay | 2 weeks postoperatively
  Number of days from the date of surgery to the date of hospital discharge, as recorded in the hospital information system (NIS-SP).
Wound Healing Status | 2 weeks postoperatively
  Clinical assessment of wound healing based on medical documentation and nursing records, including presence of wound dehiscence, delayed healing, or surgical site infection, evaluated until discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- First Department of Orthopaedic Surgery, St. Anne's University Hospital and Faculty of Medicine, Masaryk University, Brno, Czechia, Brno, Czechia, Czechia

IPD SHARING:
Plan to Share IPD: No